CLINICAL TRIAL: NCT05063071
Title: Effectiveness and Safety of Tenofovir Alafenamide for HBV Prophylaxis in Post Orthotopic Liver Transplant With HBV-related Disease
Brief Title: Tenofovir Alafenamide for HBV Prophylaxis in Post Orthotopic Liver Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAF-Prophylaxis-Post Liver Tx
Record Dates: First submitted 2021-08-18; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-07

CONDITIONS: HBV; POST LIVER TRANSPLANT
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAF monotherapy without HBIG (Experimental): The standard dose of TAF 25mg daily was used. TAF can be used on the first day after orthotopic liver transplantation. No HBIG was used before, during, or after transplantation; and therapeutic vaccination was not routinely used.
  Interventions: Drug: Tenofovir Alafenamide 25 MG

INTERVENTIONS:
Drug: Tenofovir Alafenamide 25 MG — After orthotopic liver transplant, all patients will receive Tenofovir Alafenamide monotherapy without HBIG for HBV Prophylaxis.

SUMMARY:
TAF treatment for HBV prophylaxis could lead to significant reduction in ALT and significant improvement in renal function. However, data are scarce regarding to TAF monotherapy without HBIG for HBV prophylaxis in post orthotopic liver transplant with HBV-related disease. This study is based on a real-world, multi-center, prospective study to assess the effectiveness and safety of TAF for HBV prophylaxis, which will fill in gaps with TAF monotherapy without HBIG in post liver transplant.

DETAILED DESCRIPTION:
LT has evolved rapidly, becoming the standard therapy for acute and chronic liver failure of a variety of aetiologies, with more than 80,000 procedures performed to date [13]. HBV infection is a worldwide public health problem, especially in China. The need for an antiviral treatment with NAs for liver transplant recipients has two objectives: the improvement of liver function and to decrease the risk of HBV recurrence after transplant. TAF, TDF and ETV are currently the first-line therapy in patients with CHB in all CHB treatment guidelines, which have a greater potency and higher barriers to resistance. TAF treatment for HBV prophylaxis could lead to significant reduction in ALT and significant improvement in renal function. However, data are scarce regarding to TAF monotherapy without HBIG for HBV prophylaxis in post orthotopic liver transplant with HBV-related disease. This study is based on a real-world, multi-center, prospective study to assess the effectiveness and safety of TAF for HBV prophylaxis, which will fill in gaps with TAF monotherapy without HBIG in post liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be capable of understanding and signing written informed consent; Before commencing the study procedure, participants must obtain informed consent. If the patient is hepatic Coma, the family member shall sign the written informed consent.
* ≥18 years old.
* Orthotopic liver transplant for HBV-related disease (such as HCC, DCC or liver failure). Patients were all positive for HBsAg for at least 6 months prior to liver transplantation.
* HBV DNA ≤ 2000 IU/mL before orthotopic liver transplant . (Including patients who received or did not receive oral antiviral therapy before liver transplantation)

Exclusion Criteria:

* Post OLT patients received HBIG
* Other solid organs transplant recipients
* HCV, HDV or HIV coinfection
* Other primary end-stage liver diseases (PBC, PSC, etc)
* Patients with underwent liver re-transplantation
* Liver grafts from HBsAg+ donors
* Graft dysfunction of any other causes
* HCC with primary portal vein thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-07-29 (Estimated); Study Completion 2022-12-29 (Estimated)

PRIMARY OUTCOMES:
HBV DNA undetectable rate at week 48. | 48 weeks
  evaluate the HBV DNA undetectable rate (defined as HBV DNA < 20 IU/mL) at week 48 after liver transplant.

SECONDARY OUTCOMES:
HBV DNA undetectable rate at week 96 | 96 weeks
  evaluate the HBV DNA undetectable rate (defined as HBV DNA < 20 IU/mL) at week 96 after liver transplant.
HBsAg negative rate at week 48 | 48 weeks
  evaluate the HBsAg negative rate at week 48 after liver transplant.
HBsAg negative rate at week 96 | 96 weeks
  evaluate the HBsAg negative rate at week 96 after liver transplant.
ALT normalization rate at week 48 | 48 weeks
  evaluate the ALT normalization rate at week 48 after liver transplant.
ALT normalization rate at week 96 | 96 weeks
  evaluate the ALT normalization rate at week 96 after liver transplant.
Changes in Serum Creatinine at week 48 | 48 weeks
  evaluate the change of Serum Creatinine at week 48 after liver transplant.
Changes in Serum Creatinine at week 96 | 96 weeks
  evaluate the change of Serum Creatinine at week 96 after liver transplant.
Changes in eGFR (MDRD) at week 48 | 48 weeks
  evaluate the change of eGFR (MDRD) at week 48 after liver transplant.
Changes in eGFR (MDRD) at week 96 | 96 weeks
  evaluate the change of eGFR (MDRD) at week 96 after liver transplant.
Changes in β2-MG:Cr at week 48 | 48 weeks
  evaluate the change of β2-MG:Cr at week 48 after liver transplant.
Changes in β2-MG:Cr at week 96 | 96 weeks
  evaluate the change of β2-MG:Cr at week 96 after liver transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No